CLINICAL TRIAL: NCT03959384
Title: Efficacy and Safety of Curosurf® in Patients Under 12 Months of Age Requiring Invasive Mechanical Ventilation for Acute Respiratory Distress Syndrome in the Course of Bronchiolitis: A Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Efficacy and Safety of Curosurf® in Patients Invasively Ventilated for Severe Bronchiolitis Under 12 Months of Age
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to COVID19 hospital admissions by patients with moderate-severe bronchiolitis have drastically decreased from 02/2020 to date. Moreover, many centers that had initially joined the study project had great difficulties in the activation phase
Sponsor: Azienda Ospedaliera Universitaria Integrata Verona (Other)
Responsible Party: Principal Investigator, Paolo Biban, Director, Department of Neonatal and Pediatric Critical Care, Azienda Ospedaliera Universitaria Integrata Verona
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SURFABRON
Record Dates: First submitted 2019-04-09; First posted 2019-05-22 (Actual); Last update posted 2021-04-15 (Actual); Status verified 2021-04

CONDITIONS: Bronchiolitis, Viral
MeSH Terms: conditions — Bronchiolitis, Viral | interventions — poractant alfa; Particulate Matter

STUDY DESIGN:
Intervention Model Description: multicenter, double-blind, placebo-controlled, randomized trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Patient's parents and the doctors/nurses responsible for the patient's care will be blinded. At each center only a physician and a nurse will know and prepare the drug or placebo, being subsequently not clinically involved in the care of that particular patient. The assignment of the type of treatment will be communicated by the Coordinator centre in an individual way and reserved to the researcher attending the patient's bed. The same medical researcher will then take care of administering the treatment assigned to the patient, masking the procedure with appropriate precautions. The preparation and administration of treatment can be done with the help of a nurse who does not have to disclose the type of treatment assigned. Thereafter, such a nurse will not be involved in the patient's care until the conclusion of the study. The patient evaluation will be carried out by other physicians and/or nurses who will not be aware of the type of treatment carried out.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surfactant replacement (Curosurf) (Experimental): 1. Broncho-alveolar lavage (BAL) with 25 mg / kg of Curosurf, diluted 1:10 with physiological solution, divided in two aliquots administered with a endotracheal tube in two different postures (1st BAL on right decubitus, 2nd BAL on left decubitus).
  2. Following supplementation of a dose of 25 mg / kg of Curosurf, diluted with physiological solution 1: 2 (1 ml = 40 mg of surfactant), given in two aliquots with endotracheal tube in two different postures (1st on right decubitus, 2nd on left decubitus). The treatment assigned may be repeated at least 12 hours later and in any case within 24 hours from the first treatment, at the same dosage and with the same method of administration
  Interventions: Drug: Curosurf 80Mg/Ml Intratracheal Suspension
- Ambient Air (Placebo Comparator): 1. Broncho-alveolar lavage (BAL) with air, administered with a endotracheal tube in two different postures (1st BAL on right decubitus, 2nd BAL on left decubitus).
  2. Following supplementation of air given with endotracheal tube in two different postures (1st on right decubitus, 2nd on left decubitus). The treatment assigned may be repeated at least 12 hours later and in any case within 24 hours from the first treatment, at the same dosage and with the same method of administration
  Interventions: Other: Ambient Air

INTERVENTIONS:
Drug: Curosurf 80Mg/Ml Intratracheal Suspension — CUROSURF is a natural surfactant obtained from swine lungs containing almost exclusively phospholipids, in particular phosphatidylcholine (about 70% of the total phospholipid content) and about 1% of low molecular weight hydrophobic proteins, specific for surfactant, SP-B and SP -C. CUROSURF will be administered via endotracheopulmunary.
  Other Names: phospholipid fraction from porcine lung
  Arms: Surfactant replacement (Curosurf)
Other: Ambient Air — Ambient air aspirated in sterile syringes
  Arms: Ambient Air

SUMMARY:
Background. Viral bronchiolitis is a common cause of hospitalization for acute respiratory insufficiency in young infants. Despite several RCT have tested the effectiveness of various agents, currently there is no proven specific therapy for bronchiolitis, treatment remaining mostly supportive. Based on available studies, exogenous surfactant replacement in bronchiolitis is likely to have a promising safety and efficacy profile. Primary objective. To evaluate whether Curosurf treatment is effective compared to placebo (air) in reducing the duration of invasive mechanical ventilation in the first 14 days of hospitalization, in infants less than 12 months suffering from acute hypoxemic bronchiolitis. Methods. a multicenter, double-blind, placebo-controlled, randomized trial. 19 Italian PICUs will enroll children less than12 months with hypoxemic acute bronchiolitis, with need for invasive mechanical ventilation. Once the patient has been recruited, randomization should occur as quickly as possible. The first dose of Curosurf or placebo should be administered within 60 minutes of randomization. The treatment may be repeated once, not before 12 hours and not later than 24 hours after the initial dose. The assignment of the type of treatment will be communicated by the Coordinator center to the researcher attending the patient's bed. The same medical researcher will then take care of administering the assigned treatment, masking the procedure with appropriate precautions, for example with screens or closing the patient's room whenever possible. The preparation and administration of treatment, medication or placebo, can be done by a nurse who must not disclose the assigned treatment and will not be involved in the patient's care until the conclusion of the study. Patient evaluation will be carried out by other physicians and/or nurses who will not be aware of the assigned treatment. Regardless the received treatment, all patients will be assisted according to standard practice of the Unit. For the purposes of the study, several parameters will be collected 15 minutes before, and 2, 6, 12, 24, 36, 48 hours after administration of the drug: oxygenation indexes such as OI, OSI, PaO2 and SatO2; Invasive ventilation parameters, i.e. current volume, positive end expiratory pressure, peak pressure, respiratory rate, FiO2 and mean airway pressure; and ventilation indexes such as PaCO2 and End Tidal CO2. If it is necessary to repeat the treatment, the above parameters will be re-collected with the same timepoints. During the study all the AE/ADR will be recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Aged > 40 weeks (correct gestational age) and < 12 months.
2. Patient intubated and mechanically ventilated for at least 6 hours, with expected requirement of ventilatory support of at least 24 hours.
3. Clinical picture strongly suggestive for acute bronchiolitis (fever of probable viral origin, fine crackles, prolonged expiration, lung hyperexpansion on chest X-ray)
4. Moderate or severe pediatric acute respiratory distress syndrome, defined by a Oxygenation Index (OI) > 8 or an Oxygen Saturation Index (OSI) > 7.5
5. Written informed consent obtained from both parents

Exclusion Criteria:

1. Severe prematurity (gestational age < 32 weeks). Patients with gestational age less than 32 weeks will be excluded because they are considered at high risk for respiratory pathology following their severe prematurity. This consideration does not apply in successive gestational ages. Therefore patients with mild prematurity, i.e. with gestational age equal to or greater than 32 weeks, are not to be excluded.
2. Recent phase of oxygen dependency (need for oxygen supplementation to maintain satO2 > 94% in the four weeks preceding hospitalization in Pediatric ICU)
3. Invasive mechanical ventilation for more than 24 hours.
4. Oxygenation index (OI) > 30
5. Cyanotic congenital heart disease
6. Untreated pneumothorax
7. Neuromuscular diseases
8. Severe Neurological Alterations
9. Other severe congenital anomalies
10. Indication not to attempt resuscitation
11. Patient already recruited for other clinical studies

Ages: 40 Weeks to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 9 (Actual)
Dates: Start 2019-01-09 (Actual); Primary Completion 2021-04-09 (Actual); Study Completion 2021-04-09 (Actual)

PRIMARY OUTCOMES:
Number of days free from invasive mechanical ventilation | day 14
  Number of days free from invasive mechanical ventilation within the first 14 days of hospitalization. Ventilation-free days will start after the first successful extubation (at least 48 hours without the need for re-intubation)

SECONDARY OUTCOMES:
Number of days free from non-invasive mechanical ventilation in the post-extubation phase | day 14
  Number of days free from non-invasive mechanical ventilation in the post-extubation phase
Number of cases requiring new intubation | day 14
  Number of cases requiring new intubation after previous extubation in 14 days from randomization.
Number of days of patients in PICU | day 14
  Number of days of patients in PICU
Number of days of hospitalization | day 14
  Number of days of hospitalization.
Number of days free from oxygen supplementation | day 14
  Number of days free from oxygen supplementation
Values of the Oxygen Saturation Index (OSI) | detected 15 minutes before administration of treatment and at a distance of 2, 6, 12, 24, 36 and 48 hours
  Changes in the Oxygen Saturation Index (OSI)
Values of the mechanical ventilation parameter (MAP) during invasive mechanical respiratory support | detected 15 minutes before administration of treatment and at a distance of 2, 6, 12, 24, 36 and 48 hours
  Changes in the ventilatory parameter (MAP) during invasive mechanical respiratory support
Number of patients undergoing a repeated treatment (Curosurf or placebo) | within 24 hours of the first treatment
  Number of patients undergoing a repeated treatment (Curosurf or placebo). The repetition of the assigned treatment may take place at least 12 hours apart and in any case within 24 hours of the first treatment, at the same dosage and with the same method of administration
Number of patients undergoing unconventional or more invasive treatments (HFOV, Nitric Oxide, ECMO) | during the first 14 days
  Number of patients undergoing unconventional or more invasive treatments (HFOV, Nitric Oxide, ECMO)
Rate of deaths | (1) Mortality during the first 14 days of hospitalization (2) Mortality from the date of the first intervention until the date of hospital discharge
  Rate of deaths before hospital discharge
Number of serious desaturation episodes, severe bradycardia, extreme bradycardia or cardiac arrest, pulmonary hemorrhage, pneumothorax | within the first 48 hours after treatment
  Number of serious desaturation episodes (SatO2 < 75%), episodes of severe bradycardia (FC < 80/min) , episodes of extreme bradycardia or cardiac arrest with the need for chest compressions and/or administration of drugs for resuscitation, episodes of pulmonary hemorrhage, episodes of pneumothorax

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Biban, MD, Principal Investigator — AOUI Verona
Locations (1):
- Azienda Ospedaliera Universitaria Integrata Verona, Verona, Italy

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available within 9 months of study completion, up to five years
Access Criteria: Data access request will be reviewed by the Steering committee. Requestors wil be required to sign a Data Access Agreement

REFERENCES:
- [Derived] Biban P, Conti G, Wolfler AM, Carlassara S, Gitto E, Rulli I, Moscatelli A, Micalizzi C, Savron F, Sagredini R, Genoni G, Binotti M, Caramelli F, Fae M, Pettenazzo A, Stritoni V, D'Amato L, Zito Marinosci G, Calderini E, Scalia Catenacci S, Berardi A, Torcetta F, Bonanomi E, Bonacina D, Ivani G, Santuz P. Efficacy and safety of exogenous surfactant therapy in patients under 12 months of age invasively ventilated for severe bronchiolitis (SURFABRON): protocol for a multicentre, randomised, double-blind, controlled, non-profit trial. BMJ Open. 2020 Oct 19;10(10):e038780. doi: 10.1136/bmjopen-2020-038780. PMID 33077567